CLINICAL TRIAL: NCT06844747
Title: Comparison of the Ultrasound-guided Erector Spinae Plane Block and Wound Infiltration for Postoperative Pain Management in Lumbar Disc Surgery
Brief Title: Postoperative Pain in Lumbar Disc Surgery
Acronym: Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İrem DURMUS, Principal Investigator, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023/514/250/34
Record Dates: First submitted 2025-02-12; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Erector Spinae Plane Block; Wound Infiltration; Lumbar Disc Herniation; Postoperative Pain
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The study design was double-blind, prospective, randomized, and controlled, involving patients undergoing elective lumbar disc herniation surgery.The patients were randomized into two groups, the ESPB group (Group E) and the WI group (Group W), with 25 patients in each group, using a computer system. ESPB or WI was administered to the patients according to the randomization before awakening after the operation.
Who Masked: Participant, Investigator
Masking Description: The study was initially conducted without prior registration, but a registration number is now required for publication
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- erector spinae plane block (Active Comparator): At the end of the surgery, while the patient was still intubated and in the prone position, the linear probe of a Samsung HM70 EVO ultrasound device was placed sagittally, approximately 2-3 cm lateral to the spinal cord. After identifying the erector spinae muscle and transverse processes, a 22-G, 10-mm block needle (Braun Stimuplex Ultra 360, Germany) was advanced posterior to the transverse process after reaching the bone structure. The location of the needle tip was then confirmed, 0.25% bupivacaine (20mL) was injected intermittently, and separation of the erector spinae muscle from the transverse process was observed. The procedure was applied bilaterally (22 patients)
  Interventions: Other: erector spinae plane block(ESPB)
- wound infiltration (Active Comparator): In Group W, a dose of 0.5% bupivacaine (20 ml) was injected for wound infiltration into the surgery site. (24 patients)
  Interventions: Other: erector spinae plane block(ESPB)

INTERVENTIONS:
Other: erector spinae plane block(ESPB) — ESPB group received US-guided plane block, WI group received local anaesthetic wound infiltration
  Other Names: wound infiltration

SUMMARY:
This study included 46 patients who underwent lumbar disc herniation surgery under general anesthesia. After the operation, US-guided ESPB was performed on Group E, and WI was performed on Group W. Postoperative pain was assessed, and the time to first analgesic requirement, total analgesic amount in 24 hours, and side effects were recorded. IBM SPSS Statistics 22 was used for statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologists (ASA) physical status I-II

Exclusion Criteria:

* Patients with recurrent lumbar disc herniation,
* Obesity (body mass index >35 kg/m2),
* Infection in the surgical site,
* Known local anesthetic drug allergy,
* Chronic pain, and coagulation disorders were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
US-guided ESPB and WI on postoperative pain | postoperative 1 hour, 3 hours, 12 hours, and 24 hours
  Postoperative pain assessment was conducted in the recovery unit using the Numeric Rating Scale (NRS) with a scale of 0 (no pain) to 10 (worst pain imaginable). Standard postoperative intravenous analgesia included 75 mg of diclofenac sodium administered every 8 hours. In cases where NRS was ≥4, rescue analgesia was provided with 100 mg of intravenous tramadol. Anesthesia duration, surgical duration, NRS scores at postoperative 1 hour, 3 hours, 12 hours, and 24 hours, time to first analgesic, and total analgesic requirement in the first 24 hours were recorded. All side effects (hypotension, bradycardia, etc.) were documented.

CONTACTS AND LOCATIONS:
Overall Officials: Irem DURMUS MD, Principal Investigator
Locations (1):
- Kartal Dr Lutfi Kirdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No